CLINICAL TRIAL: NCT02023151
Title: Predicting the Clinical Response to Omalizumab With Anti-IgE Response or Syk Expression in Basophils
Brief Title: Predicting the Clinical Response to Omalizumab With Anti-Immunoglobulin E (IgE) Ab Response or Syk Expression in Basophils
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00081287
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omalizumab (Other): Active
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab
  Other Names: xolair

SUMMARY:
This research is being done to test whether differences in blood cells at baseline (start of the study) can be used to predict how well omalizumab will work in a patient. Omalizumab (Xolair) is a drug approved by the U.S. Food and Drug Administration (FDA) to treat asthma. Studies show that omalizumab improves the symptoms of asthma but some people experience better improvement than others.

DETAILED DESCRIPTION:
From a therapeutic perspective, the study will determine whether changes in the peripheral blood basophil response to crosslinking anti-IgE Ab during treatment with omalizumab predicts the clinical efficacy of treatment with the drug. Secondary outcomes measures would focus on whether the starting level of anti-IgE-mediated histamine release, or the changes syk expression or its starting level would be sufficient to predict the clinical outcome.

The study is a single-site trial to evaluate the utility of baseline basophil measures to predict the efficacy of subcutaneously administered omalizumab as an add-on therapy for the treatment of adult patients 18-75 years old who have been diagnosed with moderate to severe asthma according to current approved guidelines. Patients will be treated with omalizumab according to the standard FDA approved dosing table for a period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate-to-severe asthma; male and females aged 18-75 who are symptomatic despite treatment with inhaled corticosteroids if they also had an asthma duration > 1 year.
* Positive blood testing to at least one common allergen (including must mite, D. F. and D. P., cockroach, dog or cat)
* Serum IgE within the bounds of the dosing table (>30 IU/ml to < 700 IU/ml)
* Reversibility of > 12% within 30 minutes after administration of albuterol or history of reversibility in past or history of positive methacholine in past
* Baseline Forced expiratory volume (FEV1) of > 0% and < 80% of predicted
* Treatment with 400 to 800 ug day of beclomethasone dipropionate or its equivalent.
* Patients must be willing to give written informed consent and be able to adhere to dose and visit schedules and meet trial requirements.
* Patients will be excluded if they have prior sensitivity to omalizumab, and acute respiratory tract infection prior to or during the run-in period, or a need for regular B-agonist use.

Exclusion Criteria:

* Treatment with an investigational agent within 30 days of screening
* Previously treated with omalizumab within a year prior to screening
* Treatment 1 month prior to screening with: hydroxychloroquine, methotrexate, cyclosporine, cyclophosphamide, intravenous immunoglobulin G, and plasmapheresis
* Clinically relevant laboratory anomalies at screening including individuals with reduced hematocrit (<32%), White Blood Cell (WBC) count (2400/microliter), platelet count (< 75000/microliter), and increased creatinine (> 141.4 micromolar/L), or aminotransferase (AST) (>100 IU/L).
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy, or bleeding disorder.
* History of any medical condition that is unstable
* Inability to comply with study and follow-up procedures
* Patients may not take systemic corticosteroids within 2 weeks prior to screening\
* Women of childbearing potential who are pregnant or nursing mothers, or who are of childbearing potential (post-menarche) and are not practicing an acceptable form of contraception ( as determined by the site investigator)
* Individuals with body weight less than 30 kg or greater than 150 kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarbjit S. Saini, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma & Allergy Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: Active
  Omalizumab
Period: Overall Study
Arm/Group | Omalizumab
Started | 17
Completed | 13
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Omalizumab
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Peripheral Blood Basophil Response to Crosslinking Anti-IgE Ab
Description: Data will be analyzed for the fold change in the in vitro anti-IgE-mediated histamine release response
Time Frame: baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: Fold change in basophil Syk expression
Arm/Group | Omalizumab
Number analyzed (Participants) | 13
Fold change in basophil Syk expression | 7.8 (4.8)

2. Secondary Outcome: Changes in Syk Expression
Description: Change in syk expression. Syk is a signaling molecule that is the first downstream event in IgE receptor activation of basophils.
Time Frame: baseline and 26 weeks
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Omalizumab
Number analyzed (Participants) | 13
fold change | 2.3 (.4)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Omalizumab
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=13)
Infections (Infections and infestations) | 10 (12)

LIMITATIONS AND CAVEATS:
Small study with difficult enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No